CLINICAL TRIAL: NCT01665365
Title: Long-term Clinical Outcome in Patients Undergoing Remote Ischemic Conditioning Before Primary Percutaneous Coronary Intervention for ST-elevation Myocardial Infarction: a Follow-up Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Oxford University Hospitals NHS Trust (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30685
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2013-08

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
Keywords: Myocardial infarction; Remote ischemic conditioning; Clinical outcome
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Remote ischemic perconditioning (Experimental): Intermittent arm ischemia through four cycles of 5-min inflation and 5-min deflation of a blood-pressure cuff started in the ambulance before admission to primary percutaneous coronary intervention (intervention group).
  Interventions: Procedure: Remote ischemic perconditioning
- 2. (No Intervention): Primary percutaneous coronary intervention (control group).

INTERVENTIONS:
Procedure: Remote ischemic perconditioning — Intermittent arm ischemia through four cycles of 5-min inflation and 5-min deflation of a blood-pressure cuff started in the ambulance before admission to primary percutaneous coronary intervention.
  Arms: 1. Remote ischemic perconditioning

SUMMARY:
The aim of this prospective follow-up study is to investigate 5-year clinical outcome in patients with ST-elevation myocardial infarction undergoing remote ischemic conditioning before primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain before admission to hospital within 12 h of onset, ST-segment elevation of > 0,1 mV in 2 or more contiguous leads, 18 years or older.

Exclusion Criteria:

* left bundle branch block, previous myocardial infarction, fibrinolytic treatment in the previous 30 days, previous coronary bypass surgery, left main stem stenosis requiring coronary bypass surgery, severe heart failure requiring mechanical ventilation or use of an intra-aortic balloon pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2007-02; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 5 years
  MACCE defined as all-cause mortality, readmission for heart failure, myocardial infarction, and ischemic stroke/transient ischemic attack. Data are collected from Danish nationwide registries and medical records.

SECONDARY OUTCOMES:
LV-function and remodeling | 5 years
  LV-function and remodeling measured by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid D Sloth, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Skejby, Aarhus N, Denmark